CLINICAL TRIAL: NCT01024660
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Design, Multicentre Study in Patients With Mild to Moderate Alzheimer's Disease to Investigate the Effect on Cognitive Function as Measured by Repeated CogState Testing in Relation to Effects on Traditional Cognitive Measures After 12 Weeks
Brief Title: The Effect of Cognitive Function as Measured by Repeated Cognitive Measures After 12 Weeks Treatment With Donepezil
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2285M00010
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease
Keywords: Patients with Mild to Moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 5 mg Donepezil (first 14 days), 10 mg Donepezil (next 70 days)
  Interventions: Drug: Donepezil
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo to match Aricept

INTERVENTIONS:
Drug: Donepezil — 5 mg capsule, orally, once daily, first 14 days of treatment
  Other Names: Aricept
  Arms: 1
Drug: Donepezil — 10 mg, orally, once daily, for remaining 70 days of treatment
  Other Names: Aricept
  Arms: 1
Drug: Placebo to match Aricept — Placebo capsule, orally, 84 days of treatment
  Arms: 2

SUMMARY:
The purpose of this study is to determine if there is improvement or measurable change in cognition after only one month of treatment with donepezil when using a computerized test battery. The results at one month will be compared with the results at 3 months to evaluate this.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable AD according to NINCDS-ADRDA criteria.
* The patient should live with an appropriate caregiver at home, or in a community dwelling. A caregiver should be capable of accompanying the patient to clinic visits or attending study visits in the patient's home.
* Patient and caregiver should understand, speak, and read local language.

Exclusion Criteria:

* Significant neurological disease or dementia other than AD, e.g., mixed dementia, frontotemporal dementia, and Parkinson's Disease.
* Females of child bearing potential
* Impaired vision or hearing

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
CogState Computerized Neurological Test Battery | Tl. of 25 times: 10 times between Days 3-14, 5 times between Days 36-42, 5 times between Days 64-70, four times between Days 92-97, 1 time on Day 98

SECONDARY OUTCOMES:
Neuropsychological Test Battery (NTB) | Tl. of 5 times: Once between Days 1-2, Once anytime between Days 3-14, Once anytime between Days 36-42, Once anytime between Days 64-70, Once between Days 92-97
Alzheimer Disease Assessment Scale-Cognitive (ADAS-Cog) | Tl. of 5 times: Once between Days 1-2, Once anytime between Days 3-14, Once anytime between Days 36-42, Once anytime between Days 64-70, Once between Days 92-97
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) | Tl. of 4 times: Once anytime between Days 3-14, Once anytime between Days 36-42, Once anytime between Days 64-70, Once between Days 92-97

CONTACTS AND LOCATIONS:
Overall Officials: Malene Jensen, Study Director — Study Delievery Director, AstraZeneca
Locations (18):
- Canada (5):
  - Research Site, Ottawa, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Reearch Site, Québec
- Peru (3):
  - Research Site, Callao, Lima
  - Research Site, Callao
  - Research Site, Lima
- Poland (8):
  - Research Site, Chojnice
  - Research Site, Gdansk
  - Research Site, Kalisz
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Sopot
  - Research Site, Ścinawa
  - Research Site, Warsaw
- South Africa (2):
  - Research Site, Cape Town, Western Cape
  - Research Site, Roodepoort

REFERENCES:
- [Derived] Karin A, Hannesdottir K, Jaeger J, Annas P, Segerdahl M, Karlsson P, Sjogren N, von Rosen T, Miller F. Psychometric evaluation of ADAS-Cog and NTB for measuring drug response. Acta Neurol Scand. 2014 Feb;129(2):114-22. doi: 10.1111/ane.12153. Epub 2013 Jun 13. PMID 23763450